CLINICAL TRIAL: NCT04889014
Title: Efficacy of Personal Pharmacogenomic Testing as an Educational Tool in the Pharmacy Curriculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1602413309
Record Dates: First submitted 2021-05-04; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: We investigated the effect of PGET on student knowledge, comfort, and attitudes related to pharmacogenomics (PGx) in a non-blinded, randomized controlled trial. Consenting participants were randomized to receive PGET or no PGET (NPGET) during four subsequent years of a PGx course.
Who Masked: Investigator
Masking Description: Instructors and all study personnel were blinded to participant PGET assignment, PGx results, and survey results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal genomic educational testing (PGET) (Active Comparator): PGET group participants received their own pharmacogenomic testing results prior to the course modules covering material tested in the knowledge assessment
  Interventions: Genetic: Personal genomic educational testing (PGET)
- No personal genomic educational testing (NPGET) (Placebo Comparator): No PGET (NPGET) group participants did not receive their own pharmacogenomic testing results until after study completion.
  Interventions: Genetic: No personal genomic educational testing (NPGET)

INTERVENTIONS:
Genetic: Personal genomic educational testing (PGET) — PGET consisted of a panel of pharmacogenomic variants
  Arms: Personal genomic educational testing (PGET)
Genetic: No personal genomic educational testing (NPGET) — Lack of pharmacogenomic testing
  Arms: No personal genomic educational testing (NPGET)

SUMMARY:
The purpose of this study is to evaluate the use of personal genomic educational testing (PGET) on student knowledge and clinical skills surrounding pharmacogenomic testing to ensure it is of educational benefit to our student population. Students will be provided the opportunity to opt-in to test their own pharmacogenomic panel while participating in the standard curriculum. Students will have the option of using their own reports or dummy reports during classroom activities. Our hypothesis is that those students who have their own pharmacogenomics tested will show better overall performance.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent for participation in the study
* Enrolled in 3rd year Doctor of Pharmacy course

Exclusion Criteria:

* Unwilling or unable to provide consent for participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Pharmacogenomics Knowledge Assessment | 8-12 weeks
  Improvement in performance on a knowledge assessment including eleven questions

SECONDARY OUTCOMES:
Change in Self Assessment Questionnaire | 8-12 weeks
  Improvement in Likert Scale Responses for 27 questions (scale of 1[worst] to 6[best])

IPD SHARING:
Plan to Share IPD: No